CLINICAL TRIAL: NCT03168282
Title: Evaluation of Culture Negative Severe Acute Respiratory Infection in Mexico
Acronym: CNSARI
Status: Terminated | Type: Observational
Why Stopped: Enrollment goal could not be met.
Sponsor: Mexican Emerging Infectious Diseases Clinical Research Network (Network)
Collaborators: Secretaria de Salud, Mexico (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CNSARI
Record Dates: First submitted 2017-05-04; First posted 2017-05-30 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Severe Acute Respiratory Infection (SARI)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swab; Broncho-alveolar Lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the feasibility of identifying novel etiologic agents associated with SARI in patients who have required intubation and in whom, after analysis, a causative agent was not identified by standard microbiologic (culture) and multiplex real-time Polymerase Chain Reaction (PCR) platforms. Taking into account that isolation of any pathogens is generally time sensitive, the study will evaluate subjects that are culture negative at the time of consent. Not all subjects will actually prove to be culture negative. Additionally, the study will compare etiologic agents identified on broncho-alveolar lavage (BAL) to etiologic agents identified by routine upper airway testing on all subjects with SARI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Willing to provide informed consent; or a legal representative is willing to sign informed consent;
* Intubated due to an independent clinical decision by a clinician responsible for the patient's clinical care and NOT affiliated with the research);
* Meet WHO's SARI definition (modified) - all of the criteria below:
* History of fever, subjective feverishness or measured fever of ≥ 38.0 °C, or hypothermia as defined for Systemic Inflammatory Response Syndrome (SIRS) (<36.0 °C );
* Cough or other respiratory symptoms, such as rapidly progressing dyspnea;
* Onset within the last 21 days (as long as the clinical condition is considered acute and due to the severity it requires intubation); and
* Requiring hospitalization

Exclusion Criteria:

* Intubated for reasons other than SARI (cardiovascular accident, surgery);
* Known microbiologic diagnosis of SARI or respiratory illness:
* Any contraindication to BAL by bronchoscopy as determined by the treating physician
* Bacterial culture or other microbiologic testing for underlying etiology positive would be excluded;
* In women: Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from hospitalized patients who seek medical care due to SARI at the participating sites of LaRed Network, and who meet inclusion criteria and do not meet any exclusion criteria. For those who accept participation, either personally or through a Legally Authorized Representative (per all applicable legal and regulatory requirements complying with the sites regulations) the study will be explained and informed consent will be obtained. The study population will not include children. Pregnant women are not eligible.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Presence of etiologic agents among patients with SARI and whose culture, and multiplex PCR prove to be negative. This outcome will be described as a list of etiologic agents identified as well as the percentage of the sample affected. | Baseline

SECONDARY OUTCOMES:
Results of NP multiplex real-time PCR as compared to results from samples taken from the lower respiratory tract through BAL. | Baseline
  The comparison will allow for determining difference between upper airway nasopharyngeal (NP) Multiplex real-time results and lower respiratory multiplex real-time PCR results.
Results of NP microRNA as compared to results from samples taken from the lower respiratory tract through BAL. | Baseline
  The comparison will allow for determining difference between upper airway nasopharyngeal (NP) microRNA results and lower respiratory microRNA results.
Inflammatory profile of BAL samples, that will include measure of cytokine, chemokine, and growth factor levels. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Galindo-Fraga, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Santiago Pérez Patrigeon, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (3):
- Mexico (3):
  - Hospital Central de San Luis Potosí "Dr. Ignacio Morones Prieto" (SLP)., Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ), Mexico City
  - Instituto Nacional de Enfermedades Respiratorias (INER), Mexico City

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared at the end of the study, by establishing collaborations with LaRed. Initial contact would occur through the principle investigators.